CLINICAL TRIAL: NCT05148819
Title: Assessment of Sexual Dysfunction Among COVID-19 Recovered Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Abdalla Ibrahim, Post graduate student, Assiut University
Other Study IDs: PCSD
Record Dates: First submitted 2021-12-06; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 pandemic has affected hundreds of millions globally(https ://coronavirus.jhu.edu/map.html), and hundreds of thousands in Egypt(https://www.care.gov.eg/EgyptCare/Index.aspx).

However, the long-term consequences of the disease are still largely unknown. Data from 2002-2004 epidemics of SARS suggest that cardiovascular sequelae, such as microangiopathy, cardiomyopathy and impaired endothelial function, are to be expected also in COVID-19 patients.(Vittori et al, 2020) Hyperinflammation and immunosuppression are prominently featured in COVID-19, causing a cytokine storm leading to development of micro-thrombosisand disseminated intravascular coagulation (DIC). (Jose et al, 2020).

These findings can be extremely relevant for male and female sexual health: indeed, based on these premises, there is quite enough evidence to hypothesize that consequences of COVID-19 can extend to sexual and reproductive health. (Sansone et al, 2020)

A self-administered questionnaire will be disseminated using online electronic social network (Facebook, What's App) including:

Sociodemographic age& gender. Sexual dysfunction will be assessed using International Index of Erectile Function-5 (IIEF-5) for males, and Arabic Female Sexual Function Index (ArFSFI) for females will be applied.

Covid-19 related factors.

DETAILED DESCRIPTION:
The pandemic of coronavirus disease (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) represents a first-time challenge for healthcare. Despite of social distancing and isolation measures, the number of affected patients is growing daily. (Isidori et al, 2020) As of November 14th , 2021, more than 253.2 million COVID-19 cases have been confirmed worldwide, with more than 5 million deaths& more than 229.3 million subjects have recovered from COVID-19 worldwide. (https ://coronaviru s.jhu.edu/map.html)

While in Egypt more than 343 thousand COVID-19 cases with more than 19 thousand deaths have been confirmed& more than 282 thousand recoveries. (https://www.care.gov.eg/EgyptCare/Index.aspx)

However, the long-term consequences of the disease are still largely unknown. Data from 2002-2004 epidemics of SARS suggest that cardiovascular sequelae, such as microangiopathy, cardiomyopathy and impaired endothelial function, are to be expected also in COVID-19 patients. (Vittori et al, 2020)

Hyperinflammation and immunosuppression are prominently featured in COVID-19, causing a cytokine storm leading to development of micro-thrombosisand disseminated intravascular coagulation (DIC). (Jose et al, 2020)

This cytokine storm is strongly associated with the development of interstitial pneumonia (IP), however, although lungs are the primarily targeted organs, the cardiovascular system is globally affected.(Sun X et al, 2020)

Evidence in this regard supports the notion that the exaggerated production of early response proinflammatory cytokines, increases the risk of vascular hyperpermeability,possibly progressing to multiple organ failure and,ultimately, death.(Sansone et al, 2020)

Additionally, both venous and arterial thromboembolic complications as deep venous thrombosis (DVT) and stroke, including endothelial inflammation, have been reported. (Lodigiani et al, 2020)

Indeed, a growing body of evidence seems to support the theory that the endothelium is targeted by the SARS-CoV-2; (Sardu et al, 2020) most importantly, the endothelium expresses the protein angiotensin-converting enzyme 2 (ACE2),through which the virus can access host cells. (Zhang et al, 2020)

Endothelial dysfunctions, therefore, a pivotal determinant of COVID-19symptoms. (Jung et al, 2020)

These findings can be extremely relevant for male and female sexual health: indeed, based on these premises, there is quite enough evidence to hypothesize that consequences of COVID-19 can extend to sexual and reproductive health. (Sansone et al, 2020)

There is very limited literature on the incidence of sexual dysfunctions, particularly in women.(McCabe et al, 2016)

Studies on the incidence of sexual dysfunction in women are scarce and there is a deficiency of data available on this topic. In a recent study from the United Kingdom, Burri and Spector found that 5.8% of women reported symptoms that constituted a diagnosis of Female Sexual Dysfunction(FSD) and15.5% reported lifelong FSD.

There are few epidemiologic surveys addressing the incidence,as opposed to prevalence, of sexual disorders in men and there are large differences among existing studies. These differences can be explained by variations in study design, populations studied, and definitions of sexual dysfunctions. Because of these variations, itis impossible to specify the incidence of sexual dysfunctions inmen. Most research has been conducted on Erectile Dysfunction(ED). The most important common theme of the studies is that the incidence of sexual dysfunctions increases with age. (McCabe et al, 2016)

A self-administered questionnaire will be disseminated using online electronic social network (Facebook, What's App) including:

1. Sociodemographic age& gender.
2. Sexual dysfunction will be assessed using International Index of Erectile Function-5 (IIEF-5) for males, and Arabic Female Sexual Function Index (ArFSFI) for females will be applied.
3. Covid-19 related factors:

   1. Duration of infection
   2. Fever
   3. Duration since recovery (in months)
   4. Diagnosis done by (PCR, rapid test, other)
   5. Complications (respiratory, vascular, cardiac, other)
   6. Quarantine (ICU, hospital, home, other)
   7. Positive family of positive COVID-19
   8. Spouse's sexual function
   9. Anticoagulants and antiplatelets

ELIGIBILITY:
Inclusion Criteria:

* 1. Age:

  1. Men: 18-60 years
  2. Women: 18- 50 years

     2. Marital Status: Married

     Exclusion Criteria:

     Chronic Diseases:

     Patients with known history of any chronic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Was calculated using epi info statistical package version 7. Based on the following parameters for cross sectional study; assumed sexual dysfunction proportion 0.50, acceptable margin of error 0.05, design effect 1, 95% confidence level. The required sample size will be 384 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Identification of the prevalence of sexual dysfunction among covid-19 survivors. | December 2022

SECONDARY OUTCOMES:
To evaluate and compare the duration since recovery and sexual dysfunction. 3- To evaluate and compare the duration since recovery and sexual dysfunction. 3- To evaluate and compare the duration since recovery and sexual d | December 2022

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Ismaiel, Professor, Study Director — Professor of Dermatology, Venereology and Andrology, Faculty of Medicine, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
anonymous questionnaire to evaluate the effect of COVID-19 recovered patients on their sexual function.

REFERENCES:
- [Background] Isidori AM, Pofi R, Hasenmajer V, Lenzi A, Pivonello R. Use of glucocorticoids in patients with adrenal insufficiency and COVID-19 infection. Lancet Diabetes Endocrinol. 2020 Jun;8(6):472-473. doi: 10.1016/S2213-8587(20)30149-2. Epub 2020 Apr 23. No abstract available. PMID 32334645
- [Background] Vittori A, Lerman J, Cascella M, Gomez-Morad AD, Marchetti G, Marinangeli F, Picardo SG. COVID-19 Pandemic Acute Respiratory Distress Syndrome Survivors: Pain After the Storm? Anesth Analg. 2020 Jul;131(1):117-119. doi: 10.1213/ANE.0000000000004914. No abstract available. PMID 32541584
- [Background] Jose RJ, Manuel A. COVID-19 cytokine storm: the interplay between inflammation and coagulation. Lancet Respir Med. 2020 Jun;8(6):e46-e47. doi: 10.1016/S2213-2600(20)30216-2. Epub 2020 Apr 27. No abstract available. PMID 32353251
- [Background] Sun X, Wang T, Cai D, Hu Z, Chen J, Liao H, Zhi L, Wei H, Zhang Z, Qiu Y, Wang J, Wang A. Cytokine storm intervention in the early stages of COVID-19 pneumonia. Cytokine Growth Factor Rev. 2020 Jun;53:38-42. doi: 10.1016/j.cytogfr.2020.04.002. Epub 2020 Apr 25. PMID 32360420
- [Background] Sansone A, Mollaioli D, Ciocca G, Limoncin E, Colonnello E, Vena W, Jannini EA. Addressing male sexual and reproductive health in the wake of COVID-19 outbreak. J Endocrinol Invest. 2021 Feb;44(2):223-231. doi: 10.1007/s40618-020-01350-1. Epub 2020 Jul 13. PMID 32661947
- [Background] Lodigiani C, Iapichino G, Carenzo L, Cecconi M, Ferrazzi P, Sebastian T, Kucher N, Studt JD, Sacco C, Bertuzzi A, Sandri MT, Barco S; Humanitas COVID-19 Task Force. Venous and arterial thromboembolic complications in COVID-19 patients admitted to an academic hospital in Milan, Italy. Thromb Res. 2020 Jul;191:9-14. doi: 10.1016/j.thromres.2020.04.024. Epub 2020 Apr 23. PMID 32353746